CLINICAL TRIAL: NCT05706935
Title: Evaluation of the MeMed BV® Test in Adult Emergency Department Patients With Fever and Acute Respiratory Symptoms
Brief Title: MeMed BV® Test Evaluation in Adult Emergency Department Patients
Status: Completed | Type: Observational
Sponsor: University of Wisconsin, Madison (Other)
Responsible Party: Sponsor
Other Study IDs: 2022-1612; SMPH/EMERG MED (Other: UW Madison); Protocol Version 1/13/2023 (Other: UW Madison)
Record Dates: First submitted 2023-01-20; First posted 2023-01-31 (Actual); Last update posted 2024-02-01 (Actual); Status verified 2024-01

CONDITIONS: Respiratory Infection; Respiratory Infections in Old Age; Respiratory Infection Virus; Respiratory Infection Bacterial
MeSH Terms: conditions — Respiratory Tract Infections

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: None Retained — Saliva and mouth swabs, blood samples
Oversight: FDA-regulated Drug: No | FDA-regulated Device: Yes

INTERVENTIONS:
Diagnostic Test: MeMed BV® test — The MeMed BV® test is an automated semiquantitative immunoassay that measures three nonmicrobial (host) proteins (TRAIL, IP-10, and CRP) in serum samples and is intended for use in conjunction with clinical assessments and other laboratory findings as an aid to differentiate bacterial from viral infection.

SUMMARY:
The goal of this observational study is to compare the results of a serum biomarker called the MeMed BV®, which is approved to help differentiate between bacterial and viral respiratory infections, to clinical diagnoses of adult emergency department patients presenting with recent fever and signs or symptoms of a respiratory infection. Active participation is completed during the emergency department visit and includes drawing blood, obtaining a sputum sample, and answering survey questions.

DETAILED DESCRIPTION:
The MeMed BV® is a diagnostic test newly approved by the FDA to assess the likelihood of bacterial vs. viral respiratory infections based on protein biomarkers in blood. This study aims to identify the level of agreement between the results of the MeMed BV® (bacterial/viral) and the standard of care treatment received by the participant (e.g. antibiotics for patient diagnosed with bacterial pneumonia) in order to see if implementing the MeMed BV® into standard clinical care would potentially change diagnosis.

ELIGIBILITY:
Inclusion Criteria:

* Adults presenting to the emergency department
* Subjective or objective fever within the past 7 days
* Signs or symptoms of upper or lower respiratory tract infection within the past 7 days

Exclusion Criteria:

* Prisoner
* Suspicion and/or confirmed diagnosis of infectious gastroenteritis/colitis
* Active inflammatory disease
* Congenital or acquired immune deficiency
* Chronic fungal or parasitic infection
* Infection with human immunodeficiency virus (HIV)
* Hepatitis B virus (HBV)
* Hepatitis C virus (HCV)
* Infection with active tuberculosis (TB)
* Significant trauma or burns in the last 7 days
* Patients that have undergone major surgery in the last 7 days
* Pregnancy
* Active malignancy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adults presenting to the ED with history of recent fever and signs or symptoms of acute respiratory infection.
Sampling Method: Non-Probability Sample
Enrollment: 111 (Actual)
Dates: Start 2023-02-06 (Actual); Primary Completion 2023-07-31 (Actual); Study Completion 2024-01-31 (Actual)

PRIMARY OUTCOMES:
MeMed BV® test result and diagnostic concordance | Emergency department 1 day visit
  Percent agreement between result of MeMed BV® test (bacterial or viral respiratory infection) and antibiotic prescribing by emergency medicine doctor (which implies suspected bacterial infection)

CONTACTS AND LOCATIONS:
Overall Officials: Michael Pulia, MD, PhD, Principal Investigator — University of Wisconsin, Madison
Locations (1):
- University of Wisconsin, Madison, Wisconsin, United States

IPD SHARING:
Plan to Share IPD: No

DOCUMENTS (1):
  • Informed Consent Form (2023-01-17): https://cdn.clinicaltrials.gov/large-docs/35/NCT05706935/ICF_000.pdf